CLINICAL TRIAL: NCT02723149
Title: Marijuana Approach Bias Retraining and Neural Response in Youth
Acronym: MJ-AAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 44583
Record Dates: First submitted 2016-03-14; First posted 2016-03-30 (Estimated); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Alcohol Approach/Avoidance Task; Sham Approach/Avoidance Task

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Approach Avoidance Training Condition (Experimental): The AAT group will push away the joystick from marijuana pictures 90% of the trials and pull towards the marijuana pictures 10% of the trials.
  Interventions: Behavioral: Marijuana Approach Avoidance Training
- Sham Condition (Sham Comparator): The sham group will undergo the same procedures, except the ratio for marijuana pictures will be 50% push and 50% pull.
  Interventions: Behavioral: Marijuana Approach Avoidance Training

INTERVENTIONS:
Behavioral: Marijuana Approach Avoidance Training — Approach Avoidance Training (AAT) is a novel computerized procedure that modifies implicit approach tendencies by training individuals to selectively avoid drug- related stimuli, thereby overriding habitual approach tendencies. Participants are randomized to either the treatment or sham condition. Treatment duration involves 6 training sessions of approximately 15 minutes each (400 trials). AAT requires minimal training and involves only a computer and a joystick, in which participants are either pulling or pushing the joystick when different marijuana or non-marijuana images are displayed with either yellow (pull) or blue (push) border.

SUMMARY:
This study aims to determine if a marijuana (MJ) Approach Avoidance Task (AAT) intervention reduces cannabis use compared to a control condition containing no active components of AAT. Adolescent heavy MJ users (N=40, ages 16-21) will be randomly assigned to MJ-AAT (n=20) or control condition (MJ-Sham, n=20) for three weeks. The MJ-AAT includes six sessions designed to reduce action tendencies to approach marijuana. The MJ-Sham includes six MJ-AAT-sham conditions. Substance use and cognitive assessment will identify changes in MJ use patterns and mechanisms of treatment outcomes. Additionally, using an functional magnetic resonance imaging marijuana cue reactivity task, we will determine differences in neural response in reward regions before and after 3 weeks of either AAT or sham treatment.

ELIGIBILITY:
Inclusion Criteria:

* between age 16 and 21
* having >50 lifetime marijuana use episodes and a pattern of at least weekly marijuana use for the past year (>1+/week for 52 weeks) at study entry.

Exclusion Criteria:

* not having a parent to consent (for those under age 18)
* prenatal alcohol (>2 drinks on an occasion or >4 drinks in a week) or any tobacco or illicit drug exposure
* premature birth (<34 weeks gestation), birth weight <5 lbs, or other gestational or perinatal complications
* history of a serious medical or neurological problems that could affect blood oxygen level dependent (BOLD) response, brain development, or study participation, including diabetes and recurrent migraine
* current severe Diagnostic and Statistical Manual of Mental Disorders (DSM-5) major Axis I psychiatric disorder (i.e., exclude participants with bipolar disorder, psychotic disorder)
* use of any illicit substance (e.g., cocaine, methamphetamines) other than alcohol or marijuana > 100 times
* history of major neurological disorder or head trauma (with loss of consciousness >10 minutes)
* history of learning disability, pervasive developmental disorder, or other condition requiring special education
* current use of medications that affect cerebral blood flow
* non-correctable visual or hearing problems
* non-fluent in English
* MRI contraindications (e.g., braces, claustrophobia, irremovable metal implants or piercings)
* pregnant on day of scan
* intake of psychoactive medication as tested by urine drug screen.

Ages: 16 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2015-11; Primary Completion 2016-06 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Change in marijuana use from baseline through end of intervention | From 60 days before intervention to end of 3 week intervention
  Assessing the change in marijuana use (as measured by number of days used marijuana X hits per day) from baseline to end of intervention.
Change in neural reactivity (as measured by BOLD: Blood Oxygen Level-Dependent response) in reward regions during marijuana-cue reactivity task | 3 weeks
  Assessing the change in neural reactivity to marijuana cues before and after the intervention
Change in marijuana approach tendencies (via Approach Avoidance Assessment Task) as measured by reaction times. | 3 weeks
Change in short-term marijuana use from baseline to 1 month post-intervention | From 60 days before intervention to 1 month post-intervention
  Assessing the short-term effects of intervention on marijuana use (as measured by number of days used marijuana X hits per day) from baseline to 1 month post-intervention.

SECONDARY OUTCOMES:
Change in long-term marijuana use from baseline to 1 year post-treatment | From 60 days before intervention to 1 year post-intervention
  Assessing the long-term effects of intervention on marijuana use (as measured by number of days used marijuana X hits per day) from baseline to 1 year post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay M Squeglia, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States